CLINICAL TRIAL: NCT02395757
Title: Assessment Using Microperimetry of the Risk of a Fellow Eye Progressing From Stage 3 to Stage 4 (AREDS Classification) Age-related Macular Degeneration (AMD)
Brief Title: Microperimetry and Eye Progressing From Stage 3 to Stage 4 Age-related Macular Degeneration (AMD)
Acronym: PREVISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014.862
Record Dates: First submitted 2015-02-20; First posted 2015-03-24 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2016-10

CONDITIONS: Stage 3 Age Related Macular Degeneration (AREDS Classification)
Keywords: Age Related Macular Degeneration (AMD); Microperimetry; Diagnostic
MeSH Terms: conditions — Macular Degeneration; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microperimetry (Experimental): Microperimetry exam performed in addition to the usual ophthalmological examinations for monitoring AMD.
  Interventions: Device: MAIA™ (Centervue, Padova, Italy; distributed in France by EDC Lamy, Carvin, France)

INTERVENTIONS:
Device: MAIA™ (Centervue, Padova, Italy; distributed in France by EDC Lamy, Carvin, France) — An automatic microperimetry exam of the 10° central macular coverage "expert test" (customized grid) will be performed with the MAIA™ device at each semi-annual follow-up visit.

SUMMARY:
Age-related macular degeneration (AMD) is an acquired retinal pathology affecting the central region of the retina responsible for discrimination between high spatial frequencies (reading), colour vision and the central visual field. The loss of visual acuity which occurs with the onset of AMD significantly affects patients' quality of life. In developed countries, AMD is the leading cause of vision impairment for people aged over 50 years. Its prevalence in Europe in people aged over 65 years is 3.3%. In France, around 2 million people suffer from this disease.

In the first stage of the disease it is known as age-related maculopathy (ARM). This early form of the disease can develop into intermediate AMD (stage 3 of the AREDS classification) and then advanced AMD (stage 4 AREDS), which can be atrophic or exudative. In cases of exudative AMD, the intravitreal administration of anti-VEGF drugs can limit the disease's progression.

It is therefore vital to adopt a strategy to assess the stage of the disease and provide the appropriate care management at the earliest possible stage. This is even more important for patients with advanced AMD in one eye and intermediate AMD in the fellow eye, as the risk of the fellow eye progressing to the advanced stage within 5 years is between 35% and 53%.

Microperimetry is a promising new diagnostic method which combines measurements of light sensitivity, loss of fixation and the anatomy of the retina. It offers a new approach to the functional assessment of retinal damage in patients with AMD, as it precisely correlates anatomical and functional modifications by measuring the loss of sensitivity and macular fixation. It has been shown that the more advanced the patient's AMD is, the further the parameters measured by microperimetry are from the norm.

The investigators want to assess the MAIA™ as a means of screening for AMD progression in patients with a high risk of progressing to a more advanced stage (patients presenting one eye with advanced AMD and a fellow eye with stage 3 AMD according to the AREDS classification). The research hypothesis for our proposed study is that the parameters measured using microperimetry will already show abnormal results in the study eye prior to progressing to a more advanced stage of the disease. The use of these microperimetric parameters as predictor of progression would therefore make it possible to screen eyes likely to develop from intermediate to advanced AMD at an earlier stage, and subsequently provide patients who need it with earlier follow-up, preventive treatment or adapted, personalized rehabilitation as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 50 years or over;
* Patient who has given their free, informed, signed consent;
* Patient with a French social security number or equivalent cover;
* Patient presenting one eye with stage 4 AMD (according to the AREDS classification), and drusen in the fellow eye (study eye) with at least one drusen with a diameter of over 125 microns and/or extra- foveal atrophy (stage 3 AREDS);
* Patient who is willing and able to attend all the clinical appointments required for the study and complete all the related procedures.

Exclusion Criteria:

* Patient aged under 50 years;
* Patient who refuses to take part in the study;
* Woman who is pregnant or breastfeeding;
* Protected adult as set out in French law (French Public Health Law);
* Patient presenting a study eye with stage 1, 2 or 4 AMD (AREDS classification);
* Patient presenting another maculopathy in the study eye;
* Area alteration (cornea, lens, vitreous humour) which makes it impossible to carry out and interpret the microperimetry correctly;
* Patient due to undergo cataract surgery in the study eye during the 2-year study period;
* Patients who cannot be followed up for the full 2 years;
* Patients participating simultaneously in other studies which may interfere with the study results (in either eye).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
The sensitivity of the microperimetric parameter(s) and combination(s) of parameters according to patient status at final assessment. | 24 months
  The sensitivity of the microperimetry diagnostic tool will be measured by the ratio between the number of patients presenting both positive microperimetric parameters and advanced AMD (stage 4); and the total number of patients with advanced AMD diagnosed at final assessment.

SECONDARY OUTCOMES:
The specificity of the microperimetric parameter or combination of parameters with the highest level of sensitivity | 24 months after inclusion
  The specificity of the microperimetry diagnostic tool will be measured by the ratio between the number of patients presenting both negative microperimetric parameters and no advanced AMD (stage 4); and the total number of patients with no advanced AMD diagnosed at final assessment.
The positive predictive value of the microperimetric parameter or combination of parameters with the highest level of sensitivity | 24 months after inclusion
  The positive predictive value of the microperimetry diagnostic tool will be measured by the ratio between the number of patients presenting both positive microperimetric parameters and advanced AMD (stage 4); and the total number of patients with positive microperimetric parameters.
The negative predictive value of the microperimetric parameter or combination of parameters with the highest level of sensitivity | 24 months after inclusion
  The negative predictive value of the microperimetry diagnostic tool will be measured by the ratio between the number of patients presenting both negative microperimetric parameters and no advanced AMD (stage 4); and the total number of patients with negative microperimetric parameters.
The sensitivity of the microperimetric parameters associated with the parameters from other ophthalmological examinations. | 24 months after inclusion
  The parameters of other ophthalmological examinations considered will be as follows: best corrected visual acuity measured according to ETDRS (number of letters) and Snellen scales; foveolar thickness, central 1-mm thickness, external limiting membrane (ELM) integrity, and ellipsoidal line integrity measured using SD-OCT (spectral domain optical coherence tomography). The sensitivity will be measured by the ratio between the number of patients presenting both positive parameters and advanced AMD (stage 4); and the total number of patients with advanced AMD diagnosed at final assessment.
The specificity of the microperimetric parameters associated with the parameters from other ophthalmological examinations. | 24 months after inclusion
  The parameters of other ophthalmological examinations considered will be as follows: best corrected visual acuity measured according to ETDRS (number of letters) and Snellen scales; foveolar thickness, central 1-mm thickness, external limiting membrane (ELM) integrity, and ellipsoidal line integrity measured using SD-OCT. The specificity will be measured by the ratio between the number of patients presenting both negative parameters and no advanced AMD (stage 4); and the total number of patients with no advanced AMD diagnosed at final assessment.
The sensitivity of the microperimetric parameters or combinations of parameters for the sub-group of eyes presenting reticular pseudodrusen at inclusion. | 24 months after inclusion
  The sensitivity will be measured by the ratio between the number of patients presenting both positive parameters and advanced AMD (stage 4); and the total number of patients with advanced AMD diagnosed at final assessment.
The specificity of the microperimetric parameters or combinations of parameters for the sub-group of eyes presenting reticular pseudodrusen at inclusion. | 24 months after inclusion
  The specificity will be measured by the ratio between the number of patients presenting both negative parameters and no advanced AMD (stage 4); and the total number of patients with no advanced AMD diagnosed at final assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospice Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Kodjikian L, Creuzot-Garcher C, Korobelnik JF, Tadayoni R, Delafoy I, Leal C, Bernard L, Decullier E, Huot L, Mathis T. Microperimetry to predict disease progression in eyes at high risk of age-related macular degeneration disease: The PREVISION study. Acta Ophthalmol. 2023 Mar;101(2):e135-e142. doi: 10.1111/aos.15260. Epub 2022 Sep 19. PMID 36120870